CLINICAL TRIAL: NCT06667011
Title: Impact of Implementing a Daily Learning Conversation on the Mental Well-being of Anesthesiology Teachers and Trainees
Brief Title: Feedback and Mental Well-being in Anesthesiology
Acronym: FEELING
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, DIEU Audrey, Cheffe de clinique adjointe, Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2024/18SEP/423
Record Dates: First submitted 2024-10-24; First posted 2024-10-31 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Healthy
Keywords: Imposter syndrome; Mentoring; Burnout; Feedback
MeSH Terms: conditions — imposter syndrome; Burnout, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention)
- Feedback (Experimental)
  Interventions: Behavioral: Feedback

INTERVENTIONS:
Behavioral: Feedback — learning conversation between trainee and teacher lasting 5 to 10 minutes at the end of each working day
  Arms: Feedback

SUMMARY:
The aims of the study are:

* to evaluate the mental health of anesthesia trainees and teachers in the Cliniques universitaires Saint-Luc academic hospital;
* to evaluate the effect of a daily debriefing session between trainees and teachers on the mental health of the participants at the end of a trimester;
* to identify any personal and/or institutional factors that might hinder the implementation and successful running of these debriefing sessions within our teaching hospital.

The investigators will compare the data collected by questionnaires in the "intervention" group (daily debriefing) with a control group in which no debriefing will be carried out between trainees and teachers.

DETAILED DESCRIPTION:
A recent report by the Royal College of Anaesthetists (UK) reveals that one in four qualified anesthetists is considering leaving the NHS in the next five years, resulting in over one million procedures being postponed yearly. This is a public health issue. Among the main reasons cited by these anesthetists is the negative impact they attribute to their profession on their mental health. Regarding trainee anesthetists, another report by the Royal College of Anaesthetists highlights burn-out symptoms in 85% of interns. Meanwhile, a survey of members of the European Society of Anaesthesiology and Intensive Care highlighted this year the fact that over 50% of anesthetists suffer from "imposter syndrome", first described in 1978 as the inability to internalize success and the tendency to attribute success to external causes such as luck, error or knowing the right people. This "syndrome" is more common among physicians than in the general population. It is statistically associated with burnout, anxiety, and depression.

The survey revealed that women and young anesthetists are particularly at-risk sub-groups who may preferentially benefit from targeted interventions aimed at improving their well-being. Further research is needed to explore the nature and effectiveness of such interventions.

As part of their anesthesia training, future anesthetists receive teacher feedback. This feedback, defined as communication consisting of an opportunity to comment on actions to obtain a modification or reinforcement of those actions, is not delivered in the same way by all anesthesia teachers due to a lack of training on the part of the latter, but also to a lack of standardization of practices. Yet these conversations constitute complex interpersonal exchanges in which the teacher's lack of training and the absence of a shared model between teacher and learner can be deleterious, particularly to the psychological well-being of the various parties involved.

The literature reports that trainees can sometimes perceive that the institutional culture within universities prevents honest, two-way feedback, negatively impacting the specialty's working environment and learning objectives. How relationships with faculty might influence the quality and impact of feedback delivered in future anesthetists' training is yet to be fully explored.

A learning conversation model based on the advocacy-inquiry method has been described to foster productive conversation. This methodology is adopted in the sphere of medical simulation as part of debriefing with good judgment, an approach designed to encourage open dialogue, reflection, and accurate assessment of the learner's thought process.

The determinants of this type of feedback are based on several elements. Firstly, the conversation must be non-confrontational to avoid triggering defensiveness. Secondly, the conversation must be direct and concise to maintain the participants' focus and attention, especially as these conversations occur in busy clinical environments. Thirdly, the supervisor must accurately identify trainees' knowledge gaps and teach them, avoiding appearing condescending or paternalistic by sharing concepts already known. The proper conversation will create a sense of shared ownership of a patient, emphasizing the function of both individuals as team members with a collective responsibility.

This type of feedback enables supervisors to deeply interrogate the reasons behind trainees' actions to understand their thought processes better, thus providing leverage for more in-depth teaching. This technique is not about "talking nicely" but involves the instructor increasing cooperation by making themselves vulnerable to learning and opening their opinions to questioning. Moreover, by combining this feedback with genuine curiosity, the instructor encourages exchange by respecting the trainees enough to appreciate their point of view, enhancing learning.

Psychological safety - defined as "the shared belief that the team is safe for interpersonal risk-taking, with a sense of confidence that the team will not embarrass, reject or punish someone for speaking out" - is particularly important in high-functioning clinical teams. Notably, the objective and frank nature of "advocacy-inquiry" feedback foster a culture of psychological safety by encouraging strategies associated with safe learning environments, including normalizing the discussion of mistakes, stimulating curiosity, seeking new perspectives, and recognizing the valuable contributions of all team members.

The investigators hypothesize that developing this type of conversation between teachers and trainees could promote the psychological well-being of all stakeholders involved.

The first aim of this study is to assess the mental health of trainees and anesthesia teachers working in our hospital using the Clance Impostor Phenomenon Scale (CIPS) and Maslach Burnout Inventory (MBI) scores.

The second objective is to observe whether - and to what extent - the introduction of a debriefing session in the form of a daily two-way feedback session conducted according to the principles of the "learning conversation" between teachers and trainees, over a full quarter, can influence participants' mental well-being.

The third objective is to identify any personal and/or institutional factors hindering the implementation of this learning-centered conversation method and its successful running within an academic hospital.

Data will be collected through questionnaires, which participants will complete via the secure LiveSurvey platform :

* Clance Impostor Phenomenon Scale (CIPS)
* Maslach Burnout Inventory (MBI)
* Debriefing questionnaire (Timmis & Speirs)

ELIGIBILITY:
Inclusion Criteria:

* Board-certified anesthesiologists (teachers) in the visceral, pediatric, orthopedic, or neuro-head-and-neck anesthesia areas at Cliniques Universitaires Saint-Luc.
* Anesthesia trainees assigned to the visceral, pediatric, orthopedic, and neuro-head-and-neck anesthesia departments from January 7 to April 7, 2025 at Cliniques Universitaires Saint-Luc.

Exclusion Criteria:

- None.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2024-11-04 (Actual); Primary Completion 2025-04-07 (Actual); Study Completion 2025-04-07 (Actual)

PRIMARY OUTCOMES:
Maslach Burn-out Inventory (MBI) score | up to 3 months
  A 10% improvement in the MBI score on at least one of its components (personal achievement, dehumanization, feelings of exhaustion) between the start and end of the quarter will be considered relevant.

SECONDARY OUTCOMES:
Clance Impostor Phenomenon Scale (CIPS) | up to 3 months
  A 10% reduction in the CIPS score between the beginning and end of the trimester is considered relevant.

CONTACTS AND LOCATIONS:
Locations (1):
- Cliniques universitaires Saint-Luc, Brussels, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Data will be available from the principal investigator upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: From April 2025
Access Criteria: Data will be available from the principal investigator upon reasonable request.

REFERENCES:
- [Background] Ergun S, Busse JW, Wong A. Mentorship in anesthesia: a survey of perspectives among Canadian anesthesia residents. Can J Anaesth. 2017 Apr;64(4):402-410. doi: 10.1007/s12630-017-0816-1. Epub 2017 Jan 13. PMID 28092066
- [Background] Rudolph JW, Simon R, Dufresne RL, Raemer DB. There's no such thing as "nonjudgmental" debriefing: a theory and method for debriefing with good judgment. Simul Healthc. 2006 Spring;1(1):49-55. doi: 10.1097/01266021-200600110-00006. PMID 19088574
- [Background] Timmis C, Speirs K. Student perspectives on post-simulation debriefing. Clin Teach. 2015 Dec;12(6):418-22. doi: 10.1111/tct.12369. Epub 2015 May 29. PMID 26032755
- [Background] Castillo AY, Chan JD, Lynch JB, Bryson-Cahn C. How to disagree better: utilizing advocacy-inquiry techniques to improve communication and spur behavior change. Antimicrob Steward Healthc Epidemiol. 2023 Nov 6;3(1):e201. doi: 10.1017/ash.2023.457. eCollection 2023. PMID 38028895
- [Background] Gottlieb M, Chung A, Battaglioli N, Sebok-Syer SS, Kalantari A. Impostor syndrome among physicians and physicians in training: A scoping review. Med Educ. 2020 Feb;54(2):116-124. doi: 10.1111/medu.13956. Epub 2019 Nov 6. PMID 31692028
- [Background] Vaa Stelling BE, Andersen CA, Suarez DA, Nordhues HC, Hafferty FW, Beckman TJ, Sawatsky AP. Fitting In While Standing Out: Professional Identity Formation, Imposter Syndrome, and Burnout in Early-Career Faculty Physicians. Acad Med. 2023 Apr 1;98(4):514-520. doi: 10.1097/ACM.0000000000005049. Epub 2022 Nov 1. PMID 36512808
- [Background] Ramani S, Konings KD, Mann KV, Pisarski EE, van der Vleuten CPM. About Politeness, Face, and Feedback: Exploring Resident and Faculty Perceptions of How Institutional Feedback Culture Influences Feedback Practices. Acad Med. 2018 Sep;93(9):1348-1358. doi: 10.1097/ACM.0000000000002193. PMID 29517523
- [Background] Siddiqui ZK, Church HR, Jayasuriya R, Boddice T, Tomlinson J. Educational interventions for imposter phenomenon in healthcare: a scoping review. BMC Med Educ. 2024 Jan 8;24(1):43. doi: 10.1186/s12909-023-04984-w. PMID 38191382
- [Background] Gisselbaek M, Hontoir S, Pesonen AE, Seidel L, Geniets B, Steen E, Barreto Chang OL, Saxena S. Impostor syndrome in anaesthesiology primarily affects female and junior physicians☆. Br J Anaesth. 2024 Feb;132(2):407-409. doi: 10.1016/j.bja.2023.09.025. Epub 2023 Oct 25. No abstract available. PMID 37884406